CLINICAL TRIAL: NCT05742906
Title: CorMatrix® Cor™ TRICUSPID ECM® Valve Replacement Study
Brief Title: CorMatrix Cor TRICUSPID ECM Valve Replacement - Pivotal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corvivo Cardiovascular, Inc. (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-PR-1101 Rev. L Pivotal
Record Dates: First submitted 2023-01-30; First posted 2023-02-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Tricuspid Valve Disease; Tricuspid Valve Insufficiency
Keywords: Tricuspid Valve Disease; Tricuspid Valve Dysfunction; Tricuspid Valve Regurgitation; Tricuspid Valve Replacement
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Data will be collected and reported in the following four (4) groups/cohorts:
  * Group A: Adults (≥ 21 years of age) treated with SIS 1.0 study devices
  * Group B: Pediatrics (< 21 years of age) treated with SIS 1.0 study devices
  * Group C: Adults Group A: Adults (≥ 21 years of age) treated with SIS 2.0 study devices
  * Group D: Pediatrics (< 21 years of age) treated with SIS 2.0 study devices
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Group A: Adults treated with SIS 1.0 Cor TRICUSPID ECM Valve (Other): Adults (>/= 21 years of age) treated with the SIS 1.0 Cor TRICUSPID ECM Valve
  Interventions: Device: Tricuspid valve replacement with the Cor TRICUSPID ECM Valve
- Group B: Pediatrics treated with SIS 1.0 Cor TRICUSPID ECM Valve (Other): Pediatrics (<21 years of age) treated with SIS 1.0 Cor TRICUSPID ECM Valve
  Interventions: Device: Tricuspid valve replacement with the Cor TRICUSPID ECM Valve
- Group C: Adults treated with SIS 2.0 Cor TRICUSPID ECM Valve (Other): Adults (>/= 21 years of age) treated with the SIS 2.0 Cor TRICUSPID ECM Valve
  Interventions: Device: Tricuspid valve replacement with the Cor TRICUSPID ECM Valve
- Group D: Pediatrics treated with SIS 2.0 Cor TRICUSPID ECM Valve (Other): Pediatrics (<21 years of age) treated with SIS 2.0 Cor TRICUSPID ECM Valve
  Interventions: Device: Tricuspid valve replacement with the Cor TRICUSPID ECM Valve

INTERVENTIONS:
Device: Tricuspid valve replacement with the Cor TRICUSPID ECM Valve — Tricuspid valve replacement with the Cor TRICUSPID ECM Valve for the surgical management of tricuspid valve disease or dysfunction.

SUMMARY:
The goal of this pivotal study is to demonstrate the safety and performance of the Cor TRICUSPID ECM (extracellular matrix) Valve (or Cor PEDIATRIC Tricuspid ECM Valve) for the surgical management of tricuspid valve disease and dysfunction in adult and pediatric patients. The main question(s) it aims to answer are:

* whether the device may be implanted successfully and safely, and
* whether the device effectively treats tricuspid valve disease and dysfunction through 12 months

Participants will undergo:

* preoperative evaluation
* tricuspid valve replacement with the Cor TRICUSPID ECM Valve
* postoperative evaluation, including at hospital discharge, 30 days, 6 months, and 12 months, and then annually thereafter through 5 years

DETAILED DESCRIPTION:
CorMatrix Cardiovascular, Inc. has developed a device for heart valve replacement, the Cor TRICUSPID ECM Valve for adults and the Cor PEDIATRIC Tricuspid ECM Valve for pediatrics (collectively these devices will be referred to as the Cor TRICUSPID ECM Valve(s)), which can be implanted to replace dysfunctional tricuspid heart valves. The objective of this Pivotal Study is to collect safety and effectiveness data on surgical tricuspid valve replacement procedures using the Cor TRICUSPID ECM valve to support a Humanitarian Device Exemption (HDE) marketing application.

Because the majority of tricuspid valve replacements (TVRs) (approximately 80%) are performed concomitantly with other cardiac operations, including replacements of mitral or aortic valves, it is anticipated that a portion of study subjects will require concomitant replacement or repair of a dysfunctional mitral or aortic valve, based on the clinical judgment of the investigator.

Therefore, safety with the Cor TRICUSPID ECM Valve will be established by Procedural, Technical and Device Success.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a regurgitant or absent tricuspid valve requiring surgical treatment including those patients having concomitant cardiac procedures
2. Patient/authorized legal guardian understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provides written informed consent and the pediatric patient (if applicable) provides written assent (if able) prior to procedure
3. Patient/patient's authorized legal guardian is geographically stable (or willing to return for required study follow-up) and understands and is willing to fulfill all of the expected requirements of this clinical protocol
4. Patients where the Cor TRICUSPID ECM Valve will be the physiological right-sided atrioventricular (AV) valve

Exclusion Criteria:

1. Tricuspid annulus too small (< 10mm) to accommodate the Cor TRICUSPID ECM Valve
2. Left ventricular ejection fraction (LVEF) < 25%
3. Mean pulmonary pressure ≥ 50mmHg or pulmonary vascular resistance greater than 6 Woods Units
4. Emergency cardiac procedure. An example would be a person requiring resuscitation and in cardiogenic shock. An unscheduled or unplanned emergency surgery
5. Cardiac transplant patient
6. Acute transmural myocardial infarction (MI) within 7 days of enrollment that results in cardiogenic shock
7. Patients with a single ventricle where the Cor TRICUSPID ECM Valve would be the systemic AV valve
8. Documented primary coagulopathy or uncorrected platelet disorder, including thrombocytopenia (absolute platelet count < 30k). Patient can be enrolled regardless of these parameters if in the opinion of the Investigating Surgeon the coagulopathy can be adequately reversed by transfusions. An example would be the reversal of thrombocytopenia by transfusion of platelets
9. Documented evidence of intrinsic hepatic disease (defined as liver enzyme values (aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin) that are > 5 times the upper limit of reference range within 30 days of enrollment, except in association with acute/reversible decompensation as determined by the Investigator)
10. Documented evidence of significant renal dysfunction (serum creatinine > 4.0mg/dl or GFR< 30 on the modified Schwartz formula)
11. Stroke within 30 days prior to enrollment
12. Major or progressive non-cardiac disease (liver failure, renal failure, cancer (CA)) that has a life expectancy of less than one year
13. Known cancer (cancer-free ≤ 1 year; does not include non-metastatic basal cell carcinoma or cervical carcinoma) and/or undergoing treatment including chemotherapy and radiotherapy
14. Hematological disorders (e.g., aplastic anemia) or patients taking bone marrow suppressant drugs
15. Known sensitivity to porcine materials
16. Contraindication to anticoagulation/antiplatelet therapy (aspirin (ASA) and/or Plavix)
17. Patients who are pregnant (method of assessment Investigator's discretion)
18. Patients who are currently enrolled in another investigational study or registry that would directly impact the treatment or outcome of the current study, without CorMatrix written approval

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome - Procedural Success | 30 days
  Device Success and no tricuspid valve device-related Serious Adverse Events (SAEs)
Effectiveness Outcome - Individual Patient Success | 6 months
  * Device success and
  * no Cor TRICUSPID ECM Valve-related re-hospitalizations or re-interventions of the Cor TRICUSPID ECM Valve (clinically significant: new endocarditis of the tricuspid valve [TV], recurrence of tricuspid regurgitation [TR] > moderate, or right sided heart failure [HF]) unless endocarditis is secondary to recurrent drug abuse.
  * Improvement vs. baseline in symptoms (improvement in New York Heart Association [NYHA] [adult subjects] and clinical improvement [pediatric subjects] Class >/= 1 grade)
Effectiveness Outcome - Individual Patient Success | 12 months
  * Device success and
  * no Cor TRICUSPID ECM Valve-related re-hospitalizations or re-interventions of the Cor TRICUSPID ECM Valve (clinically significant: new endocarditis of the tricuspid valve [TV], recurrence of tricuspid regurgitation [TR] > moderate, or right sided heart failure [HF]) unless endocarditis is secondary to recurrent drug abuse.
  * Improvement vs. baseline in symptoms (improvement in New York Heart Association [NYHA] [adult subjects] and clinical improvement [pediatric subjects] Class >/= 1 grade)

OTHER OUTCOMES:
Technical Success | One week or prior to hospital discharge
  * Alive at exit from OR with:
  * Successful implant of the single intended Cor TRICUSPID ECM Valve
  * No need for additional emergency surgery or re-intervention related to the Cor TRICUSPID ECM Valve device
  * Final post-op transthoracic echocardiogram (TTE) (at 1 week or prior to discharge) shows tricuspid valve regurgitation </= moderate
Device Success | 30 days
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate
Device Success | 6 months
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate
Device Success | 12 months
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate
Device Success | 24 months
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate
Device Success | 36 months
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate
Device Success | 48 months
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate
Device Success | 60 months
  No device-related mortality, with
  * Original intended Cor TRICUSPID ECM Valve in place, and
  * No additional surgical or interventional procedures related to the Cor TRICUSPID ECM Valve, and
  * Intended performance of the Cor TRICUSPID ECM Valve:
    1. No clinically significant dysfunction of the tricuspid valve: defined as TR > moderate (except patients with recurrent drug abuse)
       • This includes clinically significant: detachment of the annular or papillary muscle fixation, hemolysis, para-device complications (effects on coronary circulation, paravalvular leaks) or new endocarditis, and
    2. Expected hemodynamic performance:
       * Valve mean gradient < 6mmHg [with heart rate ≤70 bpm for age ≥ 14; no HR restrictions for those <14 years] and
       * Valve regurgitation ≤ moderate

CONTACTS AND LOCATIONS:
Overall Officials: Robert Matheny, MD, Study Director — Corvivo Cardiovascular, Inc.; Brad Solberg, MBA, Study Director — Veranex
Locations (2):
- United States (2):
  - St Francis Hospital, Indianapolis, Indiana
  - Columbia University Irving Medical Center/New York Presbyterian, New York, New York

IPD SHARING:
Plan to Share IPD: No
No.